CLINICAL TRIAL: NCT01997775
Title: A Phase II Trial to Examine the Effect of Metformin on Plasma IL-6 Level in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Metformin in Stage IV Lung Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult enrollment
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Min Yeh, MD, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-102-039
Record Dates: First submitted 2013-11-17; First posted 2013-11-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: IL-6; Metformin; Non-small cell lung cancer; Lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- METFORMIN (Experimental): For patients with stage IV lung adenocarcinoma and IL-6 level higher than 2.0 pg/ml after 2 cycles of standard treatment, metformin 500mg tid orally will be given.
  Interventions: Drug: METFORMIN

INTERVENTIONS:
Drug: METFORMIN — Participants enrolled in this study will be treated with either chemotherapy (Cisplatin 75mg/m2 plus Pemetrexed 500mg/m2 on D1) for 4 cycles or targeted therapy (Gefitinib 250mg/d) till disease progression according to physicians' decision. For participants with plasma IL-6 > 2.0 pg/mL after 2 cycles of chemotherapy or targeted therapy, Metformin 500mg orally qd will be given on Day 1 of cycle 3. If patient could tolerate it well, metformin will be titrated to 500mg bid in the following week (Cycle 3 D8) and 500mg tid in the 3rd week (Cycle 3 D15). For patients receiving chemotherapy, metformin will be used for total 12 weeks and plasma IL-6 level will be checked at the end of metformin treatment. For patients receiving targeted therapy, metformin will be used till disease progression and plasma IL-6 level will be measured after use of metformin for 12 weeks.
  Other Names: GLUCOPHAGE

SUMMARY:
The purpose of this study is to determine whether metformin is effective in lowering plasma IL-6 level and improving the treatment response in patients with non-small cell lung cancer

DETAILED DESCRIPTION:
Interleukin-6 (IL-6) plays an important role in the pathogenesis of lung cancer. Several clinical studies show metformin could decrease IL-6 level in addition to the glucose-lowering effect. Preclinical data also reveal metformin could decrease the IL-6 production in lung cancer cells and enhance cytotoxicity of chemotherapy in animal model. Based on these findings, the purpose of this study is to determine whether metformin is effective in lowering plasma IL-6 level and improving the treatment response in patients with non-small cell lung cancer clinically. Patients with stage IV lung adenocarcinoma will be enrolled in this study and receive standard treatments for lung cancer, either chemotherapy combining cisplatin and pemetrexed or targeted therapy (Gefitinib). For patients with plasma IL-6 more than 2.0 pg/ml after 2 cycles of standard treatment, metformin will be given and titrated to 1500mg/day gradually. Plasma IL-6 level will be checked after use of metformin for 12 weeks. Tumor response to the standard treatment plus metformin will be evaluated and side effects of metformin will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed lung adenocarcinoma.
2. Stage IV disease as defined by AJCC 7th edition staging.
3. At least one measurable lesion (as defined by RECIST v1.1).
4. No prior radiotherapy, chemotherapy, surgery, target therapy, or immunotherapy for NSCLC. (Except the surgery for biopsy or port-A implantation, palliative localized radiotherapy for bone metastasis).
5. Age ≤ 80 years old and ≥ 20 years old.
6. ECOG performance status of 0-2.
7. Adequate organ function, including followings

   Bone marrow:

   Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; WBC ≥ 3.0 x 10^9/L Platelet count ≥ 100 x 10^9/L Hemoglobin ≥ 9g/dL

   Hepatic:

   Total bilirubin level ≤ 1.0 x UNL AST and ALT ≤ 3.0 x UNL;

   Renal:

   Creatinine level ≤ 1.5 mg/dL in men, ≤1.4 mg/dL in women; or Estimated CCr ≥ 60 mL/min. (CCr is estimated by Cockcroft-Gault formula, as appendix II)(CCr is estimated by Cockcroft-Gault formula)
8. Estimated life expectancy of at least 6 months.
9. Written (signed) Informed Consent.

Exclusion Criteria:

1. With other primary malignancies, except those remain disease-free for 3 or more years after curative treatment, basal cell cancer of the skin or in situ cervical cancer.
2. Use of other anti-cancer therapy, including chemotherapy, target therapy, immunotherapy, radiotherapy, and hormone therapy.
3. Prior participation in any investigational drug study within 28 days.
4. Use of anti-IL-6 or IL-6-lowering agents.
5. Use of metformin in the past 6 months.
6. Poor controlled diabetes (HbA1c ≥ 8.0%).
7. Known hypersensitivity or intolerance to metformin.
8. Congestive heart failure with NYHA functional class II~IV.
9. History of lactic acidosis.
10. Significant concurrent medical diseases, such as unstable angina, acute or recent myocardial infarction (< 6 months before enrollment), COPD with frequent exacerbation, uncontrolled hypertension, or recent CVA (< 6 months before enrollment).
11. Active uncontrolled infections or HIV infection.
12. Psychiatric disorders that would compromise the patient's compliance or decision.
13. Current or planned pregnancy, or breast feeding in women.
14. Poor compliance.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The change of plasma IL-6 level after the treatment with metformin | 12 weeks

SECONDARY OUTCOMES:
The objective response rate (RR) | 2 YEARS
The progression free survival | 2 years
The overall survival | 2-years
Number of participants with adverse events | 2-years
  All adverse events (AEs) occurring after the patient receiving the first dose of study drug will be monitored and recorded. Periodic measurement of vital signs, regular laboratory evaluation for hematology and blood chemistry will be arranged and these will be graded by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grades.
Changes of quality of life | 2-years
  The quality of life will be evaluated by the EQ-5D-3L questionnaire which will be completed at baseline, during the therapy, and post-therapy period

CONTACTS AND LOCATIONS:
Overall Officials: YUMIN YEH, MD, Principal Investigator — NATIONAL CHENG-KUNG UNI. HOSP.
Locations (1):
- National Cheng-Kung Uni. Hosp., Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No